CLINICAL TRIAL: NCT03917706
Title: Development of a Quality of Life Assessment Tool for Adult Patients With a Congenital Heart Disease, Having Had Surgery During Childhood
Status: Completed | Type: Observational
Sponsor: Pierre Wauthy (Other)
Responsible Party: Sponsor-Investigator, Pierre Wauthy, Medical Director of the CHU Brugmann Hospital, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Other Study IDs: CHUB-congenital cardiopathy
Record Dates: First submitted 2018-02-08; First posted 2019-04-17 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Congenital Heart Disease: Adults suffering from congenital heart disease, followed within the CHU Brugmann hospital, operated during childhood.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Patients will be contacted by phone in order to fill in a questionnaire regarding their quality of life.

SUMMARY:
The mortality due to congenital heart diseases has decreased in recent decades, even for infants with the most complex lesions.Therapeutic advances have prolonged the lifespan of people with these diseases. However, there are specific social and psychological troubles that appear later in life and can compromise employability, insurability and social integration.

There are different types of congenital heart disease: those not operated in adulthood, and those operated for curative or palliative purposes. It is estimated that about 10 out of 1000 babies are born with a congenital cardiac malformation. One-third of these have a critical diagnosis requiring a surgical intervention.

Data from the literature show that there is an unusually high prevalence of psychosocial, neurological, developmental and psychiatric disabilities among survivors, as they enter formal education.There are many factors that influence developmental outcomes at school age. Early intervention is an essential element in controlling these comorbidities. The continuous monitoring of the development by a multidisciplinary team would make it possible to identify a developmental disorder as soon as it appears and respond to it as quickly as possible.For many children and their families, the burden of the developmental consequences is higher than the daily impact of the heart disease.

Most studies and measures of quality of life in congenital heart patients require methodological improvements.They contribute little to the scientific basis of the quality of life in these patients. Future quality of life studies must invest in rigorous conceptualization, adequate operational definition and a good measure of quality of life.

The investigators propose to develop a reproducible and reliable quality of life measurement tool, suitable for adult patients suffering from congenital heart disease and having had surgery during childhood.

ELIGIBILITY:
Inclusion Criteria:

* congenital heart disease,
* patients having had surgery during childhood,
* patients followed within the CHU Brugmann Hospital.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults suffering from congenital heart disease, having had surgery during childhood, followed within the CHU Brugmann Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Quality of life assessment | 30 minutes
  Quality of life will be assessed by means of a questionnaire adapted to adult patients suffering from congenital cardiopathy and having had surgery during childhood. There are 76 short closed questions, about 6 different domains (physical activity, social life, family life, professional life, scholarity, psychological comfort).

SECONDARY OUTCOMES:
Medical antecedents | 30 minutes
  List of medical antecedents of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Marine DENEUBOURG, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No